CLINICAL TRIAL: NCT01048177
Title: A Trial of Intravesical Therapy for Interstitial Cystitis in Patients With Generalized Vulvodynia
Acronym: VV/IC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This trial was never started
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Bruce Kahn, MD, Scripps Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-09-5381
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Vulvodynia
Keywords: vulvodynia; interstitial cystitis; pelvic pain
MeSH Terms: conditions — Vulvodynia; Cystitis, Interstitial; Pelvic Pain | interventions — Administration, Intravesical; Heparin; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Bladder instillation with heparin/ lidocaine

INTERVENTIONS:
Drug: Bladder instillation with heparin/ lidocaine — 9 bladder instillations in 6 weeks

SUMMARY:
In order to investigate whether the pain in women with vulvodynia may represent bladder origin pain, we will be performing a diagnostic test for interstitial cystitis (IC) in women with generalized vulvodynia. Those women with a positive test for IC, we will be performing a series of bladder treatments (instillations) for IC and checking symptoms throughout the trial to see if significant relief of vulvar pain can be obtained through treatment for IC.

DETAILED DESCRIPTION:
A TRIAL OF INTRAVESICAL THERAPY FOR INTERSTITIAL CYSTITIS IN PATIENTS WITH GENERALIZED VULVODYNIA

BACKGROUND:

Interstitial Cystitis (IC) is a urologic pain syndrome. The classic symptoms of IC are frequency, urgency and pain (dysuria) in the absence of an infection or other obvious source. IC has also been described as a visceral pain syndrome. In recent years, less common presentations of IC have been reported in women with primary symptoms of gynecologic pain such as endometriosis, dysparunia and vulvodynia1. This aim of this study is to further characterize the relationship between vulvodynia and IC and to see if a brief course of initial therapy for IC can relieve symptoms of generalized vulvodynia (GV)

The diagnostic criteria for IC, agreed to in the mid 1980's at an NIDDK conference, was developed for research purposes. These criteria require cystoscopy with hydrodistention in the operating room under general anesthesia. There also are multiple exclusionary criteria for diagnosis which limit its utility. The end result is that up to 60% of cases of IC can be missed using NIDDK criteria for the diagnosis of IC2. Because of these limitations, cystoscopy is now used less often for diagnosis.

In recent years, the potassium sensitivity test (PST) and the "anesthetic challenge" have been developed as alternative tests for the diagnosis of IC. These newer diagnostic techniques are less invasive and less painful than cystoscopy with hydrodistention, and are now fairly well accepted for diagnosis.

My colleagues & I first reported on a group of patients with vulvodynia who were noted to have IC as diagnosed by the PST1,3. This initial data collection was part of study of a larger group of patients with pelvic pain who were screened for urinary symptoms and tested for IC using the PST. Last month, we reported solely a series of patients presenting with GV who were tested for IC using the PST3. In this most recent report, 102 / 122 (84%) of patients with GV were found to have a positive PST. These data suggest that many patients with vulvodynia may have pain of bladder origin.

In 2008, Welk and Teichman report on a group of patients with IC treated with an alkinalized heparin-lidocaine solution instilled into the bladder (intravesical treatment) for the treatment of dysparunia 4. They found that 15/23 (65%) patients reported improvements of greater than 50% on the Patient Objective Rating of Improvement of Symptom scale. This report demonstrates that a brief course of treatment for IC can result in significant symptom relief.

Intravesical treatment of IC using a heparin-lidocaine-bicarbonate solution has become common first line treatment for many patients diagnosed with IC. Its use has been reported as part of an algorithm for the care of patients newly diagnosed with IC5. It is commonly used in conjunction with multi-modal treatment for IC, but as Welk & Teichman's paper demonstrates, it can be used alone with impressive initial results.

There are no reported head-to-head comparisons of different instillations therapies. Most instillation therapies contain heparin. Heparin is a constituent of the normal glycaso-aminoglycan (GAG) mucosal barrier in the bladder. In patients with IC, this mucosal barrier is thought to be defective, specifically with regard to the presence of heparin. The heparin is thought to "rebuild" the mucosal barrier in the bladder. Many bladder instillation therapies also contain an anesthetic such as lidocaine. The anesthetic is thought to directly treat nerves in and around the bladder through desensitization. Sodium bicarbonate acts to alkinalize the solution which has also been theorized to help with absorption or direct treatment. Lastly, we have found that some patients have had an initial burning sensation for several minutes with the concentrated three ingredient formula and that a small amount of sterile water helps to prevent this. Therefore we add the sterile water to all bladder instillations.

We believe that, in many cases, patients with vulvodynia have pain that is referred from the bladder. The next logical step in defining the relationship between vulovodynia and IC is to offer a short course of intravesical treatment for IC to patients with GV after diagnosis and observe for symptom relief. We plan to perform a potassium sensitivity test for diagnosis as we believe there is not enough published data yet to support the use of the anesthetic challenge for study purposes. We also believe that the PST can help patients with vulvodynia understand better the connection between the bladder and the vulva. Further, we are confident that the PST does not cause much discomfort as has been described in some reports. We plan to proceed with this and report our findings as described in this application. If this pilot study demonstrates significant symptom relief in this population, a placebo-control randomized trial of treatment would then be indicated. Further, if our hypothesis holds true, several treatment modalities currently used for IC could be explored for use in patients with GV. We believe that this could literally open a new door to therapy for patients with GV.

OBJECTIVE:

We plan to report the incidence of IC in a pilot group of patients with GV as detected by the PST. We also plan to report the degree of symptom relief obtained in patients with a positive PST during and after a six week course of initial intravesical therapy for IC using several validated measurement tools.

METHODS:

Patients, Study sites and IRB We plan to enroll 30-60 patients into this study. We hope to complete this study as a multi-site study with patients enrolled at two institutions. We plan to obtain IRB approval at both institutions. The enrollment period will be approximately one year from January thru December 2010.

Definition of Generalized Vulvodynia For the purposes of this report, we plan to use the definition of vulvodynia agreed upon at the 2003 meeting of the ISSVD: GV is a pain syndrome characterized by vulvar pain for at least 3-6 months duration with discomfort occurring in the absence of relevant infectious, inflammatory, or neoplastic findings and in the absence of specific clinically identifiable disorder of any kind (i.e., idiopathic). Patients with pain generally characterized as burning pain which is unprovoked, provoked or both and involving most of the vulva (not localized) will be offered enrollment. The pain can be constant or intermittent. Though intermittent symptoms are not part of the 2003 ISSVD criteria, we do plan to enroll patients with intermittent symptoms as we believe that intermittent symptoms may represent "flares" of IC. Further, patients with intermittent symptoms may have vulvodynia that had previously gone unrecognized.

Inclusion criteria We plan to enroll women 18 years or older with GV and negative tests for urine infection, negative cultures for Chlamydia and gonorrhea when indicated, and negative screens or cultures for yeast infection or bacterial vaginosis when indicated. Patient symptoms will need to include no or minimal vaginal discharge and patients will have a minimum Visual Analog Score for vulvar pain of at least 3/10.

Exclusion criteria We will exclude patients from enrollment if they use chronic narcotic pain medication or have localized vulvodynia. (We believe that localize vulvodynia is less likely of bladder origin.)

Symptom Evaluation Patients' surgical and medical histories will be reviewed and documented. A questionnaire specifically regarding symptoms or diagnoses of other pain syndromes including irritable bowel syndrome, fibromyalgia, endometriosis, chronic headaches, migraines, hyper-allergic or autoimmune disorders will be completed. Several other standardized questionnaires will also administered including: 1) Pain-Urgency-Frequency or "PUF" questionnaire, 2) O'Leary-Sant Symptom Index, 3) Short - Urinary Quality of life survey, 4) Visual analog pain scale and, 5) two days of bladder diary. A patient will be considered positive for urinary symptoms if she voids nine or more times in 24 hours or has either urgency or pain associated with the voiding process. Following the 3rd, 6th, 9th treatments, as well as 3-4 weeks following the last treatment, questionnaires will be re-administered. We plan to collect data points at multiple times during treatment as we believe that symptom relief may occur quickly. This will be useful to know in planning for subsequent studies.

Potassium Testing The PST will be performed with the patient blinded to the identity of the two solutions as previously reported.10-12. All patients and controls will receive the same information in advance of the test procedure: that two separate, unidentified solutions will be instilled in the bladder and that they will be asked to grade their reactions. In brief, 40 ml of water will be instilled into the patient's bladder for 5 minutes and any reactions of urgency or pain will be graded on a scale of 0-5 (Figure 1A). Then water will then be removed and 40 ml of a potassium solution (40 mEq KCl in 100 mL water) will be instilled and reactions similarly graded. After both solutions are instilled and removed, the patient will be asked whether one solution caused more urgency or more pain than the other. Any difference between solutions will then be graded as mild, moderate, or severe.

We will consider a PST to be positive if both of the following criteria are met: the patient's urgency or pain grade for Solution 2 was at least two points above zero, and the patient identified Solution 2 as the solution causing more symptoms. We will report results in terms of the percentage of patients with positive tests.

If neither solution is associated with any symptoms of urgency or pain, the PST will be considered negative.

If the patient reports urgency or pain associated with both solutions, the test is potentially indeterminate. Many patients with IC are both volume sensitive and solute sensitive, and when they react to both solutions, this suggests pain of bladder origin. We will rate such results as indeterminate unless Solution 2 (potassium) was more provocative of symptoms; then we will rate the test positive. The number of patients with indeterminate tests will be reported.

Bladder instillations:

Patients with a positive PST will be eligible to continue in the treatment phase of the study.

Nine bladder instillations will be performed over approximately six weeks for these patients. The solution used for bladder instillations will contain: heparin 40,000 units, lidocaine 4% - 5 ml (200 mg total dose), sodium bicarbonate 8.4 % - 3 ml and sterile water - 5 ml. This is our current standard bladder instillation therapy. For patients with a positive PST, the first bladder instillation will be performed immediately following the PST.

Study costs:

We have included the diagnosis and treatment of IC in patients with vulvodynia as a standard part of our care for patients for the past 5-7 years. Therefore, we plan to continue this as routine care and bill patients' insurance for evaluation and management services as well as bladder instillations and the PST. Our other potential study site(s) will proceed similarly. We seek the support of the National Vulvodynia Association for solely direct costs of research coordinator coverage and fellow stipend support for their work on this study. These direct costs are: Research Coordinator -10 hrs /week for 50 weeks @ 37.60 per hour including benefits = $18,800.00 plus fellow stipend support - 5 hours / week for 50 weeks @ 32.45 per hour including benefits = $8,112.50. Our total request for funding is $26,912.50.

Normally, all funds acquired for research purposes at our institution are subject to an overhead "tax" of 25-30%. Our Director of Clinical Research Development has confirmed that any NVA funds received will be applied to direct research costs and not institutional costs. Confirmation of this is available in writing under separate cover.

Future applications:

If this pilot study demonstrates significant symptom relief in patients with GV, a placebo-control randomized trial of treatment would then be indicated. Hopefully this project will lay the foundation for an application for a research grant from an institution such as the NIDDK to explore this topic further.

REFERENCES

1. Authors deleted. Am J Obstet Gynecol 2002;187:1395-400
2. Evans, R., Sant, G. Changing concepts of recognition and prevalence of interstitial cystitis Current Diagnosis of Interstitial Cystitis: An Evolving Paradigm. Urol 2007;69, Suppl,
3. Authors deleted. Gynecologic presentation of interstitial cystitis as detected by intravesical potassium sensitivity. Obstet Gynecol. 2001;98:127-132.
4. Authors deleted. Prevalence of Interstitial Cystitis in Vulvodynia Patients Detected by Bladder Potassium Sensitivity. J Sex Med. 2009 Oct; XX: XX ,
5. Welk BK, Teichman JM. Dyspareunia response in patients with interstitial cystitis treated with intravesical lidocaine, bicarbonate, and heparin. Urology. 2008 Jan;71(1):67-70.
6. Authors deleted. Management of patients with interstitial cystitis or chronic pelvic pain of bladder origin: a consensus report. Curr Med Res Opin. 2005 Apr;21(4):509-16.
7. Bachmann GA; Rosen R; Arnold LD; Burd I; Rhoads GG; Leiblum SR; Avis N SO. Chronic vulvar and other gynecologic pain: prevalence and characteristics in a self-reported survey. J Reprod Med. 2006 Jan;51(1):3-9.
8. International Society for the Study of Vulvovaginal Disease, XVII World Congress, jointly sponsored by the American College of Obstetricians and Gynecologists, October 12-16, 2003, Salvador, Brazil.
9. Moyal-Barracco, M, Lynch, PJ. 2003 ISSVD terminology and classification of vulvodynia: a historical perspective. J Reprod Med 2004; 49:772.
10. Parsons CL, Greenberger M, Gabal L, Bidair M, Barme G. The role of urinary potassium in the pathogenesis and diagnosis of interstitial cystitis. J Urol 1998;159:1862-7.
11. Parsons CL, Stein PC, Bidair M, Lebow D. Abnormal sensitivity to intravesical potassium in interstitial cystitis and radiation cystitis. Neurol Urodyn 1994;13:515 20.
12. Parsons CL. Potassium sensitivity test. Tech Urol 1996;2:171-3.

ELIGIBILITY:
Inclusion Criteria:

* We plan to enroll women 18 years or older with GV and negative tests for urine infection, negative cultures for Chlamydia and gonorrhea when indicated, and negative screens or cultures for yeast infection or bacterial vaginosis when indicated.
* Patient symptoms will need to include no or minimal vaginal discharge.
* Patients will have a minimum Visual Analog Score for vulvar pain of at least 3/10.
* In order to receive bladder instillations, patients will need to have a positive potassium sensitivity test.

Exclusion Criteria:

* We will exclude patients from enrollment if they use chronic narcotic pain medication or have localized vulvodynia. (We believe that localize vulvodynia is less likely of bladder origin).

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Reduction in pelvic pain / vulvodynia | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Kahn, M.D., Principal Investigator — Scripps Clinic
Locations (1):
- Scripps Clinic, San Diego, California, United States